CLINICAL TRIAL: NCT03498274
Title: A Comparative, Controlled, Clinical Investigation of a Currently Marketed Hearing Aid When Programmed With Two Different Fitting Methods
Brief Title: A Comparison of a Currently Marketed Hearing Aid Programmed With Two Different Fitting Methods
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient recruitmen
Sponsor: Bernafon AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: BF002-1707
Record Dates: First submitted 2018-02-28; First posted 2018-04-13 (Actual); Last update posted 2019-01-23 (Actual); Status verified 2019-01

CONDITIONS: Hearing Loss
Keywords: Fitting
MeSH Terms: conditions — Hearing Loss; Epilepsy

STUDY DESIGN:
Intervention Model Description: This is a controlled, randomized, cross-over, open label, comparative clinical investigation. A randomized cross-over design is used with half of the test subjects wearing the device fit with the traditional fitting method first and the other half using the self-directed method and then switching after approximately 10 +/-5 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fitting System (Experimental): a self-directed hearing screening based on a known algorithm from Audiology Inc. sold in an automated audiogram by Grason Stadler, GSI and a simplified version of the software. The flow of the new software is driven by the end user, but a trained professional should always assist with the fitting. The new software will first perform a hearing screening on the end user and then recommend a hearing aid and prescribe amplification to the hearing aid based on the hearing screening results.
  Interventions: Device: Fitting System
- Traditional Fitting System (Active Comparator): A traditional fitting method will be used as a control. This system is controlled by a trained professional, who performs the entire fitting without much interaction from the end user. The hearing instruments will be fit with the same settings as the experimental arm.
  Interventions: Device: Traditional Fitting System

INTERVENTIONS:
Device: Fitting System — End users will drive the screening and fitting flow; however, a trained professional is intended to assist them and help with explanations and the actual fitting of the hearing aids on the person. For a first time user the physical act of placing the hearing aid in/on the ear may create confusion. Therefore, the software is designed for an assistant to guide the user through the process and help with specific parts of the fitting or any questions in general.
  Arms: Fitting System
Device: Traditional Fitting System — The trained professional will fit the hearing aids with the traditional software that is currently used on the market. They will not involve the patient except to play demonstration tones.
  Arms: Traditional Fitting System

SUMMARY:
This study is designed to investigate the benefits of the hearing aid in the laboratory and in daily life when fitted with two different methods. Subjective and objective evaluations will be made. The aim is to show the benefits of the hearing aids with both fitting methods with the help of data obtained, and to improve the available fitting methods in order to further increase the benefit for people with hearing disorders in situations where the standard method and those trained to perform it are not available.

DETAILED DESCRIPTION:
Benefits of amplification and accessories used with it outweigh anticipated risks in mild to profound hearing impaired subjects. The basic benefit of amplification should be present with any method that the trained professional fitting the instruments uses. The goal of this study is to compare two fitting methods and determine whether the end user perceives more benefit from one fitting method over the other. The objective benefit is expected to be the same; however, the subjective benefit may be different due to a possible psychological effect from more effort or time spent by the trained professional.

Bernafon will conduct this clinical investigation to test current hearing instruments fitted with the standard procedure and a self-directed procedure. Safety and performance validation of the new self-directed fitting software is needed before release to the market.

The reason for this study is to evaluate a currently marketed, CE certified, hearing aid and determine whether different fitting methods provide the same perceived benefit. Additionally, this study will validate the safety of the fitting procedure as well as collect post market safety information about the devices themselves. The goal is to evaluate the audiological performance objectively as well as the subjective benefit. Furthermore, it is important to identify unexpected, unwanted behavior from the fitting software and the devices.

ELIGIBILITY:
Inclusion Criteria:

* All types of hearing loss (sensorineural, conductive, mixed)
* If the hearing loss is conductive or mixed it must first be approved for amplification by a physician
* All shapes of hearing loss (flat, sloping, reverse slope, notch)
* Severity ranging from mild to severe
* First time hearing aid users (never worn hearing aids before)
* German speaking
* Both genders
* Ages 18 and older
* Ability and willingness to sign the consent form

Exclusion Criteria:

* Current hearing aids users
* Contraindications for amplification
* Active ear disease
* Inability to follow the procedures of the study due to language problems, psychological disorders, dementia, or other cognitive problems of the participant
* A reduced mobility unable to attend weekly study appointments
* A reduced ability to describe auditory impressions and the usage of the hearing aids
* Uncooperative so that it is not possible to record a valid pure tone audiogram
* A strongly reduced dexterity
* With psychological problems
* Central hearing disorders
* Bernafon employees
* Family members of Bernafon employees

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2018-06-11 (Actual); Study Completion 2018-06-11 (Actual)

PRIMARY OUTCOMES:
Assessment of subjective benefit with the standardized questionnaire, International Outcome Inventory For Hearing Aids (IOI-HA) | Time frame to assess change is one month with the first measure after two weeks and the second week 3-4
  The answers to the questionnaire will be compared for each fitting method to determine if the subjective hearing aid benefit is as good when using the IMD as with the RMD. There is no numerical outcome.

SECONDARY OUTCOMES:
Assessment of speech understanding with a standardized speech test that uses the percentage of words correct to score the performance. | Time frame to assess change is one month with the first measure after two weeks and the second week 3-4
  A standardized speech test will be given after each field test to compare the two fitting methods. Percentage of correct words repeated from both fitting methods will be compared to determine whether one method helped the subjects to achieve higher speech scores.
Assessment of hearing aid preference with a questionnaire | Time frame to assess change is one month after the hearing aids have been worn with both fitting methods.
  To assess if the subjects prefer one hearing aid over the other they will complete a preference questionnaire that asks specifically which hearing aid they preferred and why. There is no point scale just a selection of Hearing aid 1 or hearing aid 2.

OTHER OUTCOMES:
Assessment of unexpected device behavior (ie. distortion) with a questionnaire | Time frame to assess change is one month with the first measure after two weeks and the second week 3-4
  To assess the system for any unexpected behaviors and to evaluate any new risk factors to ensure safety of the devices, a questionnaire that distinctly asks questions about the occurence of unexpected noises such as excessive feedback or distortion will be given to the subjects. The questionnaire is based on a 5-point scale to quantify the rate of occurrence (with 1 being never to 5 being often).

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Simon, Principal Investigator — Employee
Locations (2):
- Switzerland (2):
  - Audika, Thun, Canton of Bern
  - Audika, Bern

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cox RM, Stephens D, Kramer SE. Translations of the International Outcome inventory for Hearing Aids (IOI-HA). Int J Audiol. 2002 Jan;41(1):3-26. doi: 10.3109/14992020209101307. No abstract available. PMID 12467365

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/74/NCT03498274/SAP_000.pdf
  • Study Protocol (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/74/NCT03498274/Prot_001.pdf